CLINICAL TRIAL: NCT04295811
Title: A Multicenter Case-Control Study of the Efficacy of EsoGuard on Samples Collected Using EsoCheck, Versus Esophagogastroduodenoscopy, for the Diagnosis of Barrett's Esophagus With and Without Dysplasia, and for Esophageal Adenocarcinoma
Brief Title: Efficacy of EsoGuard Assay on Esophageal Surface Cells Collected With EsoCheck vs EGD for the Diagnosis of BE or EAC
Acronym: ESOGUARDBE2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lucid Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Organization: PAVmed Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PR-0138 / EG-CL-102
Record Dates: First submitted 2020-02-29; First posted 2020-03-05 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Barrett Esophagus; Esophageal Adenocarcinoma; Barretts Esophagus With Dysplasia; Barrett's Esophagus Without Dysplasia
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Intervention Model Description: Multi-center, single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- EsoCheck and EsoGuard vs. EGD with or without biopsies (Experimental): All subjects will undergo both the EsoGuard lab assay run on distal esophageal cells collected with EsoCheck (non-invasive esophageal cell sample collection) device followed by Esophagogastroduodenoscopy (EGD) with or without biopsies
  Interventions: Device: EsoGuard (lab assay); Diagnostic Test: Esophagogastroduodenoscopy

INTERVENTIONS:
Device: EsoGuard (lab assay) — EsoGuard assay (LDT) will be used on cells collected using the EsoCheck (510K cleared esophageal cell collection device)
  Other Names: EsoCheck (esophageal cell sample collection device)
Diagnostic Test: Esophagogastroduodenoscopy — Planned EGD to diagnose and/or treat disorders of esophagus, stomach, and small intestine. When abnormal tissues are noted, biopsies of the tissue are taken through the scope to diagnose tissue abnormalities.
  Other Names: EGD

SUMMARY:
The study will assess the performance of the combined system, i.e., the use of the EsoGuard assay (lab developed test) on cells collected using the EsoCheck (501k cleared device) to detect Barrett's Esophagus (BE), with or without dysplasia, and esophageal adenocarcinoma (EAC) as compared to Esophagogastroduodenoscopy (EGD) plus biopsies in both confirmed cases of BE/EAC and in controls (subjects without a prior diagnosis but undergoing screening for BE/EAC)

DETAILED DESCRIPTION:
This is a two phase multicenter study to assess the operating characteristics of the EsoGuard diagnostic assay panel performed on esophageal mucosal cells collected using the EsoCheck cell collection device in known "Cases" of disease (i.e., patients with a history of Barrett's Esophagus (BE) with and without varying degrees of dysplasia or intramucosal adenocarcinoma [IMC]) and in patients with no known history of these conditions. The latter are presumed to be "Controls", though this final determination is made as part of study conduct, not at the time of enrollment.

The study is divided into a Run-In phase and an Efficacy phase. The assignment of a patient to one or the other of these two phases will be made based on two pieces of information: 1) the Final Study Diagnosis (as defined below) and 2) the current tally versus the pre-determined target number of patients already assigned to each of the subgroups (e.g., non-dysplastic Barrett's Esophagus (NDBE), high grade dysplasia {HGD]) for each phase. Patients will first be enrolled into the Run-In phase subgroups. Only once the targeted enrollment for a given Run-In phase subgroup has been reached, subsequent patients with a particular diagnosis will be assigned to the appropriate Efficacy Phase subgroup, until the targeted total number is reached. Run In phase data will be maintained in a separate database from Efficacy phase data. Study conduct is identical in both phases; however, data from each phase will be segregated and analysis of each phase will be used solely for its predetermined purpose without any co-mingling of data. Once assigned, no patient, or their data, will be re-assigned or moved from being a Run-In phase patient to being an Efficacy phase patient, or from the Run-In phase database to the Efficacy phase database, or vice versa.

The Run-In phase will enroll the initial 60 short segment NDBE (also known as short segment Barrett's Esophagus [SSBE]) and 25 long segment NDBE (also known as long segment Barrett's Esophagus [LSBE]) Cases, the initial 10 low grade dysplasia [LGD] Cases, the initial 3 high grade dysplasia [HGD] Cases, and the initial 2 intramucosal adenocarcinoma [IMC] Cases, as well as the initial 100 Controls. The Efficacy phase will enroll 54 Cases each with a Final Study Diagnosis of NDBE, LGD, HGD, and IMC, and 54 Controls.

Run-In phase data will be used solely to derive the optimal numerical cutoffs by which to score mVIM and mCCNA1 (which are two genes where the methylated DNA changes are located) positivity or negativity. These cutoffs serve as the key inputs into an algorithm by which an overall EsoGuard result of positive versus negative is determined. The setting of these cutoffs will be done by Sponsor personnel with full access to all Run-In phase data; the goal will be to optimize overall EsoGuard assay sensitivity and specificity for its intended use as a screening test in the at-risk population. The assay, once validated and locked, will be used to analyze patients' distal esophageal cells obtained in both the Efficacy phase of this Case Control study as well as in a separate Screening study (PR-1039/EG-CL-101) to be conducted in parallel. Only Run-In phase data will be used to set cutoffs. The mVIM and mCCNA1 (i.e., genes with methylated DNA changes) cutoffs will be set and then the EsoGuard assay re validated and "locked", all before any Efficacy phase distal esophageal cells specimens collected from study patients will undergo EsoGuard analysis.

Sponsor personnel will have open access to all Run-In phase data during the enrollment of the Run-In phase in order to determine if the data from patients enrolled to date is sufficient to inform adequately the setting of cutoffs. If Sponsor so determines, it may elect to terminate enrollment in the Run-In phase early (i.e., prior to enrolling the 100 Cases and 100 Controls listed above). If early termination of the Run-In phase is elected, all patients enrolled subsequent to the date Sponsor makes this election will be entered into the Efficacy phase and such subsequent patients will count towards the Efficacy phase enrollment objectives.

As well, should Sponsor complete the intended Run-In phase enrollment of 100 Cases and 100 Controls but determine, upon its assessment of the resulting data, that data from additional Cases could improve the setting of cutoffs, Sponsor may decide to enroll up to 100 additional Run-In phase Cases. These 100 Cases may be in whatever distribution of disease Sponsor elects (i.e., ranging from NDBE through to IMC). In order to augment the Run-In phase patient counts, the Sponsor will set updated targets for enrollment of each Run-In phase subgroup and will assign patients to each Run-In subgroup to be augmented, based on patients' Final Study Diagnosis and on whether the updated subgroup target has been met. When each updated subgroup enrollment target has once again been met, subsequent patients with that subgroup diagnosis will be enrolled into the Efficacy phase.

ELIGIBILITY:
Inclusion Criteria:

All Patients:

1. Men aged 50 years and above
2. ≥5 years either of

   * Gastroesophageal Reflux Disease (GERD) symptoms,
   * GERD treated with proton pump inhibitor (PPI) therapy (whether symptom control is achieved or not), or
   * any combination of treated and untreated periods, as long the cumulative total is at least 5 years
3. No solid foods eaten for at least 2 hours prior to EsoCheck procedure
4. One or more of the following:

   * Caucasian race
   * Current or past history of cigarette smoking
   * Body mass index (BMI) of at least 30 kg/m2
   * First-degree relative with Barrett's Esophagus (BE) or Esophageal Adenocarcinoma (EAC)

Cases:

1. Previous diagnosis of non-dysplastic Barrett's Esophagus (NDBE), low grade dysplasia (LGD), high grade dysplasia (HGD), and/or intramucosal adenocarcinoma (IMC)
2. Diagnosis by esophagogastroduodenoscopy (EGD) (with exception of NDBE) was within 4 months prior to study enrollment
3. Indicated for surveillance EGD or for therapeutic EGD
4. Able to provide, by day of study EGD, the original glass slide(s) of biopsy specimens from most recent prior EGD

Exclusion Criteria:

1. Inability to provide written informed consent
2. On anti-coagulant drug(s) that cannot be temporarily discontinued
3. Known history of esophageal varices or esophageal stricture
4. Any contraindication, as deemed in Investigator's medical judgment, to undergoing the EsoCheck procedure, undergoing the EGD procedure, and/or having biopsies taken, including but not limited to due to comorbidities such as coagulopathy or a known history of esophageal diverticula, esophageal fistula, and/or esophageal ulceration
5. History of difficulty swallowing (dysphagia) or painful swallowing (odynophagia), including swallowing pills
6. Oropharyngeal tumor
7. History of esophageal or gastric surgery, with exception of uncomplicated surgical fundoplication procedure
8. History of myocardial infarction or cerebrovascular accident within past 6 months
9. Any known lesion which, in the opinion of the endoscopist, obstructs greater than 25% of the esophageal lumen
10. Prior participation in PR-0139/EG-CL-101 (Lucid BE Screening Study)
11. Prior EGD during which a therapeutic procedure such as, but not limited to, ablation, cryotherapy or endoscopic mucosal resection, was performed for the treatment of BE and/or EAC
12. History of esophageal motility disorder
13. Currently implanted Linx device

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 470 (Estimated)
Dates: Start 2020-06-18 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy | Per subject analysis through study completion which is up to approximately 5 weeks
  The primary efficacy endpoint is the sensitivity of EsoGuard. The primary efficacy objectives of this study are to measure the sensitivities of EsoGuard-based diagnosis in 54 cases each of non-dysplastic Barrett's Esophagus (NDBE), low grade dysplasia (LGD), high grade dysplasia (HGD), and intramucosal adenocarcinoma (IMC) in order to assess EsoGuard's ability to detect disease across the entire continuum of disease progression.

SECONDARY OUTCOMES:
Secondary Efficacy | Per subject through study completion which is up to approximately 5 weeks
  The secondary efficacy outcome will be the specificity of EsoGuard (which are run on samples collected using EsoCheck) for Controls. Specificity of EsoGuard will be calculated for the controls as the number of controls who test negative via EsoGuard divided by the total number of controls.

OTHER OUTCOMES:
Safety outcome of EsoCheck Device (510k cleared, non-invasive, esophageal cell collection device) on all patients who undergo the device procedure. | Per subject through study completion which is up to approximately 5 weeks
  Assessed by evaluation of esophageal abrasions (as visualized during esophagogastroduodenoscopy[EGD]) when EsoCheck and EGD procedures are performed the same day as well as adverse events (AEs) serious adverse events (SAEs), adverse device effects (ADEs), serious adverse devices effects (SADEs), unanticipated serious adverse device effects (USADEs) and Medical Device Deficiency Incidents.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle McDermott, Study Director — Lucid Diagnostics, Inc.
Locations (36):
- United States (30):
  - Lucid Investigative Site, Birmingham, Alabama
  - Lucid Investigative Site, Orange, California
  - Lucid Investigative Site, Aurora, Colorado
  - Lucid Investigative Site, Englewood, Colorado
  - Lucid Investigative Site, Washington D.C., District of Columbia
  - Lucid Investigative Site, Jacksonville, Florida
  - Lucid Investigative Site, Chicago, Illinois
  - Lucid Investigative Site, Shreveport, Louisiana
  - Lucid Investigative Site, Baltimore, Maryland
  - Lucid Investigative Site, Boston, Massachusetts
  - Lucid Investigative Site, Ann Arbor, Michigan
  - Lucid Investigative Site, Flowood, Mississippi
  - Lucid Investigative Site, St Louis, Missouri
  - Lucid Investigative Site, Omaha, Nebraska
  - Lucid Investigative Site, Lebanon, New Hampshire
  - Lucid Investigative Site, New Hyde Park, New York
  - Lucid Investigative Site, Rochester, New York
  - Lucid Investigative Site, Chapel Hill, North Carolina
  - Lucid Investigative Site, Portland, Oregon
  - Lucid Investigative Site, Philadelphia, Pennsylvania
  - Lucid Investigative Site, Providence, Rhode Island
  - Lucid Investigative Site, Charleston, South Carolina
  - Lucid Investigative Site, Greenville, South Carolina
  - Lucid Investigative Site, Knoxville, Tennessee
  - Lucid Investigative Site, Nashville, Tennessee
  - Lucid Investigative Site, Austin, Texas
  - Lucid Investigative Site, Dallas, Texas
  - Lucid Investigative Site, Houston, Texas
  - Lucid Investigative Site, Salt Lake City, Utah
  - Lucid Investigative Site, Richmond, Virginia
- Netherlands (6):
  - Lucid Investigative Site, Amsterdam
  - Lucid Investigative Site, Eindhoven
  - Lucid Investigative Site, Groningen
  - Lucid Investigative Site, Nieuwegein
  - Lucid Investigative Site, Nijmegen
  - Lucid Investigative Site, Rotterdam

IPD SHARING:
Plan to Share IPD: No